CLINICAL TRIAL: NCT00631800
Title: Phase II Randomized, Double Blind, Placebo Controlled, Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity Study in VLBW Neonates of BSYX-A110, for the Prevention of Staphylococcal Infection
Brief Title: Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity Study in VLBW Neonates of BSYX-A110
Acronym: N003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biosynexus Incorporated (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Gerald Fischer, MD, President and CEO, Biosynexus Incorporated
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MAB-N003
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2008-03-10 (Estimated); Status verified 2008-02

CONDITIONS: Staphylococcal Sepsis
Keywords: Staphylococcal; Monoclonal antibodies; Very Low Birth Weight Infants; Prophylaxis
MeSH Terms: interventions — pagibaximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Pagibaximab (formerly BSYX-A110)
- 60 mg/kg (Experimental): 60 mg/kg was given on Days 0, 7, 14
  Interventions: Drug: Pagibaximab (formerly BSYX-A110)
- 90 mg/kg (Experimental): 90 mg/kg was given on Days 0, 7, 14
  Interventions: Drug: Pagibaximab (formerly BSYX-A110)

INTERVENTIONS:
Drug: Pagibaximab (formerly BSYX-A110) — Pagibaximab at 60, 90 mg/kg intravenously at Days 0, 7, 14
  Other Names: BSYX-A110; HU96-110; Pagibaximab

SUMMARY:
The purpose of this study is to evaluate the safety (including tolerability), pharmacokinetics, pharmacodynamics and clinical activity of BSYX-A110 administered in a 3-dose regimen on Study Days 0, 7, and 14.

DETAILED DESCRIPTION:
This Phase II study will be a randomized, double blind, placebo controlled study of BSYX-A110 in very low birth weight neonates. A total of 80 infants will be dosed in this study. Participants will receive either BSYX-A110 or placebo, at 60 mg/kg or 90 mg/kg. The Study Drug will be administered at 48-120 hours of life, 7 days after the initial dose, and 14 days after the initial dose for all dose groups.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria at the time of first infusion (Day 0):

1. 48-120 hours of age, inclusive
2. Birth weight of 700-1300 grams
3. Inpatient in a Neonatal Intensive Care Unit
4. Written informed consent obtained from the parent(s) or legal guardian

Multiple gestations:

1. Siblings from multiple gestations may be enrolled if they each meet the entry criteria
2. No more than 4 subjects in any birth weight cohort may be siblings

Exclusion Criteria:

Patients may have none of the following at the first dose:

1. Survival not expected for at least 1 week after infusion
2. Clinically overt systemic infection, as determined by history, physical examination, and positive culture from a normally sterile site. (Infuse only when infant clinically stable and cultures negative for 48 hours. If being evaluated for sepsis, decision to infuse may be deferred as allowed by protocol infusion window. Infusions outside of protocol window must be approved by Sponsor.)
3. Severe congenital anomalies or genetic disorders that are likely to be fatal or that may interfere with drug distribution or metabolism, as determined by history and/or physical examination, and including but not limited to:

   i. Trisomy 13 ii. Trisomy 18 iii. Hypoplastic Left Heart Syndrome iv. Omphalocele v. Gastroschesis vi. Holoprosencephaly
4. Known or suspected hepatic or renal insufficiency
5. Clinically uncontrolled seizures
6. Immunodeficiency other than due to prematurity
7. A history of standard immune globulin administration prior to first study drug infusion (excluding Hepatitis B Immune Globulin, HBIG)
8. Any history, in the infant subject or its mother, of a hypersensitivity or severe vasomotor reaction to immunoglobulin G, or blood products
9. Currently receiving, recently received, or planned to receive other investigational agents that could interfere with conduct or results of this study; including enrollment in another investigational study for a product under an IRB-approved protocol
10. Expectation that the patient will not be able to be followed for the duration of the study
11. Mother with serology positive for hepatitis B surface antigen

Ages: 48 Hours to 120 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2003-05; Primary Completion 2004-03 (Actual); Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Safety and pharmacokinetics | 0 - 56 days

SECONDARY OUTCOMES:
Pharmacodynamics, sepsis/bloodstream infection | 0 - 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Weisman, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital/Ben Taub Hospital (Baylor College of Medicine), Houston, Texas, United States

REFERENCES:
- [Derived] Weisman LE, Thackray HM, Steinhorn RH, Walsh WF, Lassiter HA, Dhanireddy R, Brozanski BS, Palmer KG, Trautman MS, Escobedo M, Meissner HC, Sasidharan P, Fretz J, Kokai-Kun JF, Kramer WG, Fischer GW, Mond JJ. A randomized study of a monoclonal antibody (pagibaximab) to prevent staphylococcal sepsis. Pediatrics. 2011 Aug;128(2):271-9. doi: 10.1542/peds.2010-3081. Epub 2011 Jul 25. PMID 21788224
- See also: Biosynexus Incorporated — http://www.biosynexus.com